CLINICAL TRIAL: NCT02410733
Title: Clinical First-in-human Dose Escalation Study Evaluating the Safety and Tolerability of Intravenous Administration of a Tetravalent RNA-lipoplex Cancer Vaccine Targeting the Tumor-associated Antigens NY-ESO-1, Tyrosinase, MAGE-A3, and TPTE in Patients With Advanced Melanoma
Brief Title: Evaluation of the Safety and Tolerability of i.v. Administration of a Cancer Vaccine in Patients With Advanced Melanoma
Acronym: Lipo-MERIT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RB_0003-01; 2013-001646-33 (EudraCT Number)
Record Dates: First submitted 2015-03-24; First posted 2015-04-08 (Estimated); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Melanoma
Keywords: melanoma; Lipo-MERIT; cancer vaccine; RB_0003-01; BioNTech; BioNTech SE; BioNTech RNA; RNA; RNA vaccine; BNT111
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lipo-MERIT (Experimental): 7 dose escalation cohorts (3 +3 design) and 3 expanded cohorts
  Interventions: Biological: Lipo-MERIT

INTERVENTIONS:
Biological: Lipo-MERIT — vaccination

SUMMARY:
The purpose of this study is to determine the safety and tolerability of intravenous administration of a tetravalent RNA-lipoplex cancer vaccine targeting four tumor-associated antigens in patients with advanced melanoma.

DETAILED DESCRIPTION:
* The Lipo-MERIT vaccine consists of four naked ribonucleic acid (RNA)-drug products (DPs) that are optimized to induce antigen-specific cluster of differentiation (CD)8+ and CD4+ T cell responses against the four selected malignant melanoma-associated antigens New York-ESO 1 (NY-ESO-1), tyrosinase, Melanoma-associated antigen A3 (MAGE-A3), and Trans-membrane phosphatase with tensin homology (TPTE).
* In this study, naked RNA DPs were formulated with liposomes to form RNA-lipoplexes (RNA-LPX) that (i) protect RNA from degradation in the serum, (ii) enable in vivo targeting of antigen-presenting cells (APC), and therefore (iii) constitute a novel vaccine formulation that supports intravenous administration. As of August 31, 2021 the RNA-DPs RBL001.1, RBL002.2, RBL003.1 and RBL004.1 initially used for treatment have been replaced by the improved RNA drug substances RBL001.3, RBL002.4, RBL003.3 and RBL004.3. These drug substances are formulated in lipoplexes to yield RNA-LPX (drug product). The added maximum duration of trial treatment with the new drug products is 18 months.
* The Lipo-MERIT vaccine is expected to lead to several effects contributing to its immunological (therapeutic) effect. First, the RNA-LPX home to APCs in lymphoid organs after intravenous injection, where they are rapidly taken up by professional APCs. Incorporated RNA is translocated to the cytoplasm leading to its translation by the host ribosome complex into four Antigen encoding proteins which are processed and presented on both Human leukocyte antigen (HLA)-class I as well as HLA-class II molecules. Consecutively, antigen-specific CD8+ and CD4+ T cell responses will be triggered by HLA-peptide complexes on the surface of antigen-presenting cells.
* In addition, the Lipo-MERIT vaccine is expected to transiently activate APCs (change of surface marker expression and cytokine secretion) via signaling of Toll-like receptor (TLR)s, subsequently leading to the transient induction of inflammatory cytokines (such as Interferon (IFN)-α and Interferon gamma induced protein 10 [IP-10]) supporting the induction of tumor-antigen specific T cell responses.

ELIGIBILITY:
Inclusion Criteria:

* Cohort I: stage IV malignant melanoma (American joint committee on cancer (AJCC) 2009 melanoma classification)
* Cohorts II-VII and expanded cohorts: stage IIIB-C, or stage IV of malignant melanoma (AJCC 2009 melanoma classification) [only applicable until approval of protocol version 10.0] Expanded cohort C only patients with stage IV melanoma (AJCC 2009 melanoma classification) with measurable disease (at least one target lesion according irRECIST) [applicable for all patients included after approval of protocol version 10.0 and higher] and with disease progression at the time of first treatment with Investigational medicinal product (IMP) [applicable for all patients included after approval of protocol version 11.0]
* Therapy only for subjects not eligible or declining any other available approved therapy after all available treatment options have been transparently disclosed (to be documented!)
* Expression of either NY-ESO-1, tyrosinase, MAGE-A3, and/or TPTE confirmed by RT-qPCR analysis from formalin-fixed paraffin-embedded (FFPE)
* ≥ 18 years of age
* Written informed consent
* Eastern cooperative oncology group (ECOG) performance status (PS) 0-1
* Life expectancy ≥ 6 months
* White blood cell (WBC) ≥ 3x10^9/L
* Hemoglobin ≥ 9 g/dL
* Platelet count ≥ 100,000/mm^3
* Alanine aminotransferase/Aspartate aminotransferase (ALT/AST) < 3 x upper limit of normal (ULN) (except patients with liver metastasis)
* Negative pregnancy test (measured by Human chorionic gonadotropin [β-HCG]) for females with childbearing age

Exclusion Criteria:

* Pregnancy or breastfeeding
* Primary ocular melanoma
* Concurrence of a second malignancy other than squamous or basal cell carcinoma, non-active prostate cancer, or cervical carcinoma in situ or non-active treated urothelial carcinoma
* Brain metastases

  * Patients with history of treated or inactive brain metastasis are eligible for treatment in expanded cohort C, provided they meet all of the following criteria:
  * measurable disease outside of the brain (in addition to inactive brain metastasis);
  * no ongoing requirement of corticosteroids as therapy for brain metastases,
  * with corticosteroids discontinued ≥1 week prior to visit 2 (day 1) with no ongoing symptoms attributable to brain metastasis;
  * the screening brain radiographic imaging is ≥ 4 weeks since completion of radiotherapy
* Post-splenectomy Patients
* Known hypersensitivity to the active substance or to any of the excipients
* A serious local infection (e.g. cellulitis, abscess) or systemic infection (e.g. pneumonia, septicemia) which requires systemic antibiotic treatment within 2 weeks prior to the first dose of study medication
* Positive test for acute or chronic active hepatitis B or C infection
* Clinically relevant active autoimmune disease
* Systemic immune suppression:

  * Human immunodeficiency virus (HIV) disease
  * Use of chronic oral or systemic steroid medication (topical or inhalational steroids are permitted)
  * Other clinical relevant systemic immune suppression
* Symptomatic congestive heart failure (NYHA 3 or 4)
* Unstable angina pectoris
* Radiotherapy and minor surgery within 14 days prior to the first study treatment administration
* Myelosuppressive chemotherapy within 14 days and after reconstitution of blood values prior to the first study treatment administration
* Ipilimumab within 28 days prior to the first study treatment administration
* Treatments with BRAF inhibitors, MEK inhibitors, or the combination of both, and anti-programmed death-1 (PD-1) antibodies within 14 days prior to the first administration of study treatment (not applicable for patients with parallel treatment in expanded cohorts A, B, or C at the discretion of the investigator)
* Interferon, major surgery, vaccination, and other investigational agents within 28 days or 5 half-lives depending on what gives the longer range before the first treatment
* Approved BRAF inhibitors vemurafenib or dabrafenib, approved anti-PD-1 inhibitors nivolumab or pembrolizumab as well as approved MEK inhibitor trametinib, or the approved combination of BRAF-MEK inhibitors in patients in dose escalation cohorts. Concomitant treatment with approved BRAF inhibitors, approved anti-PD-1 antibodies or MEK inhibitor as well as the approved combination of BRAF-MEK inhibitors is allowed for patients included in the expanded cohorts, after analysis of safety data collected for the dose escalation cohorts and data and safety monitoring board (DSMB) approval. Local radiation will be allowed as concurrent treatment for patients in expanded cohort as well.

  - After approval of protocol version 10.0 and higher only anti-PD-1 antibodies are allowed for treatment of patients in expanded cohort C.
* Fertile males and females who are unwilling to use a highly effective method of birth control (less than 1% per year, e.g. condom with spermicide, diaphragm with spermicide, birth control pills, injections, patches or intrauterine device) during study treatment and for at least 28 days (male patients) and 90 days (female patients of childbearing potential) after the last dose of study treatment
* Presence of a severe concurrent illness or other condition (e.g. psychological, family, sociological, or geographical circumstances) that does not permit adequate follow-up and compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events as a Measure of safety and tolerability | up to 8 years
  Number of patients with adverse events, total number of adverse events, dose limiting toxicities

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 8 years
  ORR defined as the number of patients with complete responses (CR) or partial responses (PR) as best overall response according to Immune-related Response Evaluation Criteria in Solid Tumors criteria (irRECIST) divided by the number of patients in the efficacy analysis set.
Disease control rate (DCR) | up to 8 years
  DCR defined as the number of patients with CR or PR or stable disease (SD) as best overall response according to irRECIST divided by the number of patients in the efficacy analysis set.
Duration of response (DoR) | up to 8 years
  DoR defined as the time from initial response until first objective tumor progression according to irRECIST.
Progression Free Survival (PFS) | up to 8 years
  PFS defined as the time from the first vaccination to confirmed occurence of Progression or death from any course, which ever occurs first, per irRECIST.
Overall survival (OS) | up to 8 years
  OS defined as the time of first trial treatment until death from any cause.
Change of induced T-cell responses for Lipo-MERIT vaccine from visit 2 (day 1) to day 71 (assessed by immunoassays) | up to 8 years
  Vaccine induced T-cell responses assessed by immunoassays in skin.

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (4):
- Germany (4):
  - Johann Wolfgang Goethe Universität Frankfurt, Klinik für Dermatologie, Venerologie und Allergologie, Frankfurt
  - Universität Heidelberg, Dermatologie und NCT, Heidelberg
  - Universitätsmedizin Mainz, Hautklinik und Poliklinik, Mainz
  - Universitätsmedizin Mannheim, Klinik für Dermatologie, Venerologie und Allergologie, Mannheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sahin U, Oehm P, Derhovanessian E, Jabulowsky RA, Vormehr M, Gold M, Maurus D, Schwarck-Kokarakis D, Kuhn AN, Omokoko T, Kranz LM, Diken M, Kreiter S, Haas H, Attig S, Rae R, Cuk K, Kemmer-Bruck A, Breitkreuz A, Tolliver C, Caspar J, Quinkhardt J, Hebich L, Stein M, Hohberger A, Vogler I, Liebig I, Renken S, Sikorski J, Leierer M, Muller V, Mitzel-Rink H, Miederer M, Huber C, Grabbe S, Utikal J, Pinter A, Kaufmann R, Hassel JC, Loquai C, Tureci O. An RNA vaccine drives immunity in checkpoint-inhibitor-treated melanoma. Nature. 2020 Sep;585(7823):107-112. doi: 10.1038/s41586-020-2537-9. Epub 2020 Jul 29. PMID 32728218